CLINICAL TRIAL: NCT02765607
Title: Circulatory Oscillations in Post Cardiac Surgery Patients
Status: Completed | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/2019
Record Dates: First submitted 2016-04-19; First posted 2016-05-06 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Coronary Disease
Keywords: Blood circulation; Cardiac surgical procedures; Homeostasis
MeSH Terms: conditions — Coronary Disease | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Heart surgery

SUMMARY:
In this observational study investigators examine the presence of circulatory oscillations in blood pressure, heart rate, and doppler laser flow before and after planned cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for routine coronary artery bypass graft (CABG) surgery, single procedure only

Exclusion Criteria:

* no sinus or pacemaker rhythm
* ejection fraction below 0.5
* serious valvular disease
* right ventricular failure
* pulmonary hypertension
* serious postoperative bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for routine coronary artery bypass graft (CABG) surgery.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Frequency and amplitude of oscillations of electrocardiogram (ECG) | First day
  analyzed by continuous wavelet transform

CONTACTS AND LOCATIONS:
Overall Officials: Nils K Skjaervold, PhD, Principal Investigator — Trondheim University Hospital
Locations (1):
- Trondheim University Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No